CLINICAL TRIAL: NCT07298330
Title: A Randomized, Open-label, Multicenter, Phase 3 Trial Evaluating Brelovitug vs Delayed Treatment for the Treatment of Chronic Hepatitis Delta Infection (AZURE-4)
Brief Title: A Trial Evaluating Brelovitug vs Delayed Treatment for the Treatment of Chronic Hepatitis Delta Infection (AZURE-4)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bluejay Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJT-778-304; 2025-522105-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Chronic Hepatitis D Infection
Keywords: Hepatitis Delta virus; HDV; Hepatitis D infection; Hepatitis D virus
MeSH Terms: conditions — Hepatitis D | interventions — Treatment Delay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brelovitug 300 mg (Experimental): Participants will receive treatment with brelovitug 300 mg once weekly for 96 weeks
  Interventions: Drug: Brelovitug 300 mg
- Brelovitug 900 mg (Experimental): Participants will receive treatment with brelovitug 900 mg once every 4 weeks with a loading dose at Week 2 for 96 weeks
  Interventions: Drug: Brelovitug 900 mg
- Delayed treatment with brelovitug 300 mg (Active Comparator): Participants will have 12 weeks of delayed treatment followed by brelovitug 300 mg once weekly for 96 weeks
  Interventions: Drug: Delayed Treatment with Brelovitug 300mg

INTERVENTIONS:
Drug: Brelovitug 300 mg — Route of administration- Subcutaneous Injection
  Other Names: BJT-778; BTG
  Arms: Brelovitug 300 mg
Drug: Brelovitug 900 mg — Route of administration- Subcutaneous Injection
  Other Names: BJT-778; BTG
  Arms: Brelovitug 900 mg
Drug: Delayed Treatment with Brelovitug 300mg — Route of administration- Subcutaneous Injection
  Other Names: BJT-778; BTG
  Arms: Delayed treatment with brelovitug 300 mg

SUMMARY:
This is a Phase 3, global, randomized, open-label, multicenter trial designed to evaluate the safety and efficacy of chronic treatment with brelovitug (BJT-778) for chronic hepatitis delta virus (HDV) infection. The objective of this study is to test the safety and effectiveness of brelovitug compared to delayed treatment.

DETAILED DESCRIPTION:
The study consists of 3 study arms. Approximately 80 participants will be randomized 2:1:1 to one of the following treatment arms:

Arm 1: Participants will receive brelovitug 300 mg subcutaneously once weekly for 96 weeks.

Arm 2: Participants will receive brelovitug 900 mg subcutaneously once every 4 weeks for 96 weeks.

Arm 3: Participants will attend study clinic visits and delay treatment with brelovitug for 12 weeks. At Week 12, participants will receive brelovitug 300 mg subcutaneously once weekly for 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Chronic HDV infection
3. HDV RNA >500 IU/mL at Screening
4. ALT >ULN at Screening
5. Willing to take or already taking HBV nucleos(t)ide therapy.

Exclusion Criteria:

1. Pregnant or nursing females
2. Unwilling to comply with contraception requirements during the study
3. Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy
4. Clinical hepatic decompensation (i.e., ascites, encephalopathy variceal hemorrhage).
5. Solid organ or bone marrow transplantation
6. Presence of other liver disease(s) (non-HBV/HDV), such as metabolic dysfunction-associated steatohepatitis (MASH), alcohol associated hepatitis, cholestatic liver disease, hepatocellular carcinoma.

Note - Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a composite endpoint of virologic response and ALT normalization at Week 24 in brelovitug arms compared to response at Week 12 of delayed-treatment arm | Week 24
  The composite endpoint is defined as virologic response (HDV RNA ≥2 log10 IU/mL decrease from Baseline or undetectable HDV RNA (< the lower limit of quantification [LLOQ], target not detected [TND]) and ALT normalization (decrease in ALT from baseline to ≤ upper limit of normal [ULN])

SECONDARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events (TEAEs) | Up to 96 weeks
  An AE is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at Screening (e.g., medical history), worsens during the study (post-Baseline/ Day 1), regardless of the suspected cause of the event.
Percentage of participants who discontinue treatment due to an adverse event (AE) | Up to 96 weeks
  An AE is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at Screening (e.g., medical history), worsens during the study (post-Baseline/ Day 1), regardless of the suspected cause of the event.
Percentage of participants with HDV RNA ≥ 2 log10 IU/mL decline from baseline or TND | Up to 96 Weeks
Percentage of participants with HDV RNA <LLOQ | Up to 96 Weeks
Percentage of participants with HDV RNA <LLOQ, TND | Up to 96 Weeks
Percentage of participants with ALT normalization | Up to 96 Weeks
  ALT normalization is defined as a decrease in ALT from baseline to ≤ ULN
Percentage of participants with ALT normalization in combination with virologic response of HDV RNA ≥ 2 log10 IU/mL decline from baseline or <LLOQ, TND | Up to 96 Weeks
  The composite of participants with ALT normalization (decrease in ALT from baseline to ≤ ULN) and virologic response of HDV RNA ≥ 2 log10 IU/mL decline from baseline or TND.
Percentage of participants with ALT normalization in combination with HDV RNA <LLOQ | Up to 96 Weeks
  The composite of participants with ALT normalization (decrease in ALT from baseline to ≤ ULN) and virologic response of HDV RNA <LLOQ
Percentage of participants with ALT normalization in combination with HDV RNA <LLOQ, TND | Up to 96 Weeks
  The composite of participants with ALT normalization (decrease in ALT from baseline to ≤ ULN) and virologic response of HDV RNA <LLOQ, TND.
Percentage of participants with HDV RNA <LLOQ, TND at post-treatment follow up. | Post-Treatment Weeks 24 and 48
Change from baseline in liver stiffness as determined by transient elastography (e.g., FibroScan) | Up to 96 Weeks
Change from baseline in APRI (AST-to-platelet ratio index) | Up to 96 Weeks
Change from baseline in CTP score in participants with cirrhosis | Up to 96 Weeks
Change from baseline in Model for End-Stage Liver Disease (MELD) score in participants with cirrhosis | Up to 96 Weeks
Percentage of participants with clinical disease progression from baseline in HDV-associated liver disease. | Up to 96 Weeks
  Liver disease progression will be determined by the Independent Data Monitoring Committee (IDMC).

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - University of California, Davis, Davis, California
  - Quest Clinical Research, San Francisco, California
  - Alliance Clinical, Las Vegas, Las Vegas, Nevada
  - Prime Clinical Research Inc, Mansfield, Texas
- Georgia (4):
  - Hospital Service LTD, Kutaisi
  - Diakori LLC, Tbilisi
  - JSC T. Tsertsvadze Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LTD Academician Vakhtang Bochorishvili Clinic, Tbilisi
- Soroka University Medical Center, Beersheba, Israel
- Aga Khan University & Hospital, Karachi, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No